CLINICAL TRIAL: NCT07286201
Title: A Multicenter, Randomized, Controlled Study to Evaluate the Safety and Effectiveness of a Bioresorbable Nasal Dressing Containing Mometasone Furoate Compared to a Steroid-eluting Sinus Stent
Brief Title: Evaluation of the Safety and Performance of a Bioresorbable Nasal Dressing Containing Mometasone Furoate (MF)
Acronym: ENHANCE II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polyganics BV (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIP-6
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Rhinosinusitis (CRS); Chronic Rhinosinusitis (CRS) With and Without Nasal Polyps
Keywords: Nasal Packing; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- OCEAN (Experimental): Application after nasal/sinus surgery
  Interventions: Device: OCEAN
- Steroid-eluting Sinus Stent (Active Comparator): Application after nasal/sinus surgery
  Interventions: Device: Steroid-eluting sinus stent

INTERVENTIONS:
Device: OCEAN — Biodegradable nasal dressing applied after sinus/nasal surgery
  Arms: OCEAN
Device: Steroid-eluting sinus stent — Applied after sinus/nasal surgery
  Arms: Steroid-eluting Sinus Stent

SUMMARY:
The primary objective of the study is to evaluate the safety and effectiveness of OCEAN as an adjunct aid in wound healing after nasal/sinus surgery and to demonstrate that OCEAN is non-inferior compared to a steroid-eluting sinus stent.

DETAILED DESCRIPTION:
A multicenter, randomized, single-blinded, controlled, intra-patient non-inferiority study enrolling 110 subjects at up to 13 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject is scheduled to undergo bilateral endoscopic sinus surgery for Chronic Rhinosinusitus with nasal polyps (CRSwNP) or without nasal polyps (CRSsNP) and is indicated for bilateral complete ethmoidectomy (anterior and posterior ethmoidectomy) at a minimum. Additional sinuses may be operated on at the surgeon's discretion.
3. Subject is willing and able to provide informed consent.
4. Subject is willing and able to comply with the investigational plan requirements.
5. Subjects with a pre-operative Lund-MacKay stage of 6 (≥3 per nostril).
6. Subject with a pre-operative Lund-Mackay stage side-to-side difference ≤ 2.
7. Subject of child-bearing potential is not pregnant and agrees to not become pregnant during the course of the study.

Exclusion Criteria:

1. Subject with a history of chronic epistaxis or experienced a significant epistaxis event (defined as epistaxis requiring medical intervention) in the past 3 months.
2. Subject with an underlying systemic disorders known to affect the nose (e.g., Wegener's granulomatosis, sarcoidosis, Churg-Strauss syndrome, or other systemic vasculitides).
3. Subject with any bleeding disorder or use of medication increasing bleeding risk, except low-dose aspirin.
4. Subject with a known or suspected allergy to device components.
5. Subject with known hemophilia.
6. Subject with insulin dependent diabetes.
7. Subject with an oral steroid dependent condition.
8. Subject with glaucoma, ocular hypertension, posterior subcapsular cataracts.
9. Subject with a (previous) diagnosis of Samter's Triad (AERD).
10. Subject that requires nasal ointments or creams at time of device placement.
11. Subject with a neurological, medical, psychiatric condition, or social circumstance that would potentially increase risk, interfere with study participation, or confound interpretation of study data.
12. Subject with plans to (or otherwise anticipate the need to) undergo an ENT procedure within the 90-day study follow-up.
13. Subject participating in another clinical research study (within 30 days prior to screening up to 90 days post-operative).
14. Subject that used any form of biologics within 90 days prior to sinus surgery and during follow-up to day 25.
15. Subject that used any form of corticosteroid within 2 weeks prior to sinus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Serious Adverse Events | Up to Day 25
  Rate of serious adverse events related to the use of OCEAN bioresorbable nasal dressing.
Endoscopic Assessment | Day 25
  Endoscopic assessment of wound healing to compare test-treated and control-treated cavities.

SECONDARY OUTCOMES:
Rate of Adverse Events | Up to Day 90
  Assessment of all adverse events.
Endoscopic Evaluation of Sinonasal Cavities | Days 25 and 90
  Endoscopic evaluation of sinonasal cavities for to evaluate wound healing.
Rate of post-operative interventions | Up to Day 25 and Day 90
  Rate of post-operative interventions, including surgical intervention to separate adhesions, and/or oral steroid intervention, and/or biologics.

IPD SHARING:
Plan to Share IPD: No